CLINICAL TRIAL: NCT06787131
Title: A Double-Blind, Placebo-Controlled, First-in-Human Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ZE50-0134 in Healthy Volunteers
Brief Title: Clinical Study Aiming to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Administration of ZE50-0134 at 5 Dose Levels in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lomond Therapeutics Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ZE50-0134-0001
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Chronic lymphocytic leukemia; refractory chronic lymphocytic leukaemia; relapsed chronic lymphocytic leukaemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — Rabeprazole; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Level 1 Single dose (Experimental): Dose level 1: 6 participants will receive 100 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 2 Single dose (Experimental): Dose level 2: 6 participants will receive 200 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 3 Single dose (Experimental): Dose level 3: 6 participants will receive 400 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 4 Single dose (Experimental): Dose level 4: 6 participants will receive 800 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 5 Single dose (Experimental): Dose level 5: 6 participants will receive 1600 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 1 Single dose optional (Experimental): Dose level 1: 6 participants will receive 100 mg ZE50-0134 and 2 participants will receive placebo under fed conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 2 Single dose optional (Experimental): Dose level 2: 6 participants will receive 200 mg ZE50-0134 and 2 participants will receive placebo under fed conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 3 Single dose optional (Experimental): Dose level 3: 6 participants will receive 400 mg ZE50-0134 and 2 participants will receive placebo under fed conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 4 Single dose optional (Experimental): Dose level 4: 6 participants will receive 800 mg ZE50-0134 and 2 participants will receive placebo under fed conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 5 Single dose optional (Experimental): Dose level 5: 6 participants will receive 1600 mg ZE50-0134 and 2 participants will receive placebo under fed conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 2 Single dose + itraconazole (Experimental): Dose level 2: 6 participants will receive 200 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions (to be administered in conjunction with itraconazole [200 mg itraconazole to be administered twice per day [BID] on Day -4 and once per day [QD] on Days -3 to 8, inclusive)
  Interventions: Drug: ZE50-0134 or placebo; Drug: Itraconazole (200 mg)
- Level 3 BID dosing (Experimental): Dose level 3 BID dosing: 6 participants will receive 400 mg of ZE50-0134 administered BID and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE50-0134 or placebo
- Level 3 Single dose + Rabeprazole (Experimental): Dose level 3: 6 participants will receive 400 mg ZE50-0134 and 2 participants will receive placebo under fasted conditions (to be administered in conjunction with rabeprazole [rabeprazole 20 mg once daily (QD) on Day 1 and Day 2]).
  Interventions: Drug: ZE50-0134 or placebo; Drug: Rabeprazole 20 mg

INTERVENTIONS:
Drug: ZE50-0134 or placebo — The patients will receive ZE50-0134 or placebo.
Drug: Rabeprazole 20 mg — Rabeprazole 20 mg once daily (QD) on Day 1 and Day 2.
  Arms: Level 3 Single dose + Rabeprazole
Drug: Itraconazole (200 mg) — Itraconazole 200 mg twice per day.
  Arms: Level 2 Single dose + itraconazole

SUMMARY:
A first-in-human study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple ascending doses of ZE50-0134 administered orally in healthy volunteers.

DETAILED DESCRIPTION:
This is a double-blind, randomised, placebo-controlled study evaluating the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of a single administration of ZE50-0134 at 5 dose levels. The effect of food on ZE50-0134 may also be evaluated at each dose level (optional). The effects of CYP3A4 inhibition will also be evaluated in a single cohort. Evaluation of dose levels will be conducted in a sequential fashion with lower dose levels evaluated first in the sequence.

In this study, healthy volunteers will be enrolled to receive single ascending doses of ZE50-0134 or placebo under fasted or fed conditions. ZE50-0134 will also be evaluated in conjunction with itraconazole, to evaluate the potential effects of CYP3A4 inhibition. The starting dose will be 100 mg with 5 dose levels planned.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50.0 kg (males) or 45.0 kg (females) at screening.
4. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the screening visit and prior to dosing at the timepoints indicated in the Schedule of Assessments, including:

   1. Physical examination without any clinically significant findings.
   2. Systolic blood pressure in the range of 90 mm Hg to 160 mm Hg; diastolic blood pressure in the range of 40 mm Hg to 95 mm Hg.
   3. Heart rate (HR) in the range of 40 to 100 bpm after 5 minutes in a supine or semi-supine position
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.7°C (inclusive).
   5. No clinically significant findings in serum chemistry, hematology, coagulation and urinalysis tests as judged by the Investigator, including the following specific findings:

   i. Hemoglobin and platelet count within normal ranges (as per local laboratory standard ranges), WBC count (> 3.0 x 109/L), lymphocyte count (> 1.0 x 109/L), and neutrophil count (> 1.5 x 109/L) ii. AST, ALT and total bilirubin < 1.5 x ULN (note: for participants with Gilbert's syndrome, ULN is considered to be 2.9 mg/ml).

   iii. Additional inclusion criterion for cohort evaluating effect of CYP3A4 inhibition only: ALT, AST, ALP and gamma-glutamyltransferase (GGT) must be normal (within reference range).

   f. Triplicate 12-lead ECG (taken after the volunteer has been supine/semi-supine for at least 10 minutes) with average QTcF ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities.
5. Female volunteers must:

   1. Be of nonchildbearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause, and a follicle-stimulating hormone (FSH) level >40 IU/L at the screening visit), or
   2. If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception from signing the consent form until at least 30 days after the last dose of the study drug.
6. Male volunteers must agree not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception from signing the consent form until at least 90 days after the last dose of study drug.
7. Have suitable venous access for blood sampling.
8. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant. Note: participants with a history of fully resolved childhood asthma are permitted.
2. Acute infections within 4 weeks prior to Day -1 (nominal Cohorts 1-10) or Day -4 (nominal Cohort 11), or current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
3. Presence or history of any abnormality or illness, including gastrointestinal surgery, which in the opinion of the PI may affect absorption, distribution, metabolism or elimination of the study drug. Note: participants with Gilbert's syndrome may be permitted, at the discretion of the PI (or delegate). Participants with a history of cholecystectomy may be permitted at the discretion of the PI (or delegate).
4. Any history of malignant disease in the last 5 years (excludes surgically resected skin squamous cell or basal cell carcinoma)
5. Any screening laboratory result outside the normal laboratory reference range (as confirmed upon repeated testing) and deemed clinically significant by the PI.
6. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
7. Use of or plans to use systemic immunosuppressive (e.g., corticosteroids by any route, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 5 half-lives of individual agent or within 28 days (whichever is longer) prior to first study drug administration.
8. Use of or plans to use agents (e.g., grapefruit and grapefruit products) that have clinically significant interaction with CYP3A4 or the use of any medications that could have a significantly impact on organ function (e.g., barbiturates, omeprazole, cimetidine) during the study or within 5 half-lives of individual agent or within 28 days (whichever is longer) prior to first study drug administration. Note: timeframe = 3 days for grapefruit and grapefruit products or other foods/drinks (e.g. pomelo) that may have a clinically significant interaction with CYP3A4.
9. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or clinically significant arrythmia.
10. Participant is planning to have surgery between Screening and the EoS visit.
11. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or tuberculosis (TB) at the screening visit.
12. History of latent or active TB infection, or signs or symptoms suggestive of active TB infection upon medical history and/or physical examination.
13. Estimated creatinine clearance < 60 mL/min using the Cockcroft-Gault formula.
14. History of any drug or alcohol abuse in the past 2 years defined as >21 units of alcohol per week for males and >14 units of alcohol per week for females. Where 1 unit = 360 mL of beer, 150 mL wine, or 30 mL of spirits.
15. History of alcohol consumption in the 4 days prior to dosing.
16. Positive drugs of abuse, or alcohol breath test results at the screening visit, Day -4 prior to itraconazole administration (nominal Cohort 11 only), or at check-in (Day -1).
17. Volunteer smokes more than 5 cigarettes or equivalent per week, and/or volunteer is unwilling to abstain from smoking (including use of all tobacco products or nicotine-containing products, and smoking cessation aids such as gum or patches) for 72 hours prior to Day -4 (nominal Cohort 11 only) or check-in on Day -1 and throughout the confinement period at the study site.
18. Use of any prescription medications within 14 days or at least 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, including use of any over-the-counter medication (including herbal products, nutritional supplements, diet aids, vitamin supplements, minerals and hormone supplements) within 7 days or at least 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, with the exception of oral contraceptives and the occasional use of paracetamol (doses of 500 mg up to every 6 hours or 2 g per day maximum for no more than 3 consecutive days in one week).
19. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
20. Known hypersensitivity to any of the study drug ingredients.
21. Use of any inactivated vaccinations within 14 days, or any live vaccinations within 30 days prior to the first study drug administration.
22. For women of childbearing potential, a positive serum pregnancy test at the screening visit or a positive urine pregnancy test (with confirmatory serum pregnancy test) on Day -4 prior to itraconazole administration (nominal Cohort 11 only), or at check-in (Day -1).
23. Females who are breastfeeding or planning to breast feed at any time during the study.
24. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.
25. Receiving an investigational drug in another clinical trial within 30 days or 5 half-lives of the investigational agent (whichever is longer) prior to the first study drug administration.
26. Any other condition or prior therapy that in the opinion of the Investigators would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
27. Any history of long COVID infection (defined by continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation).

    Additional exclusion criteria for cohort evaluating the effect of CYP3A4 inhibition only:
28. History or presence of clinically significant hypersensitivity or idiosyncratic reaction to itraconazole or other azole compounds, or any inactive ingredients.
29. History or presence of clinically significant liver disease.
30. Creatinine kinase > 1.5 x ULN at screening or on Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics of ZE50-0134 | Within 15 min prior to dosing with ZE50-0134/placebo to 168 hours post-dose
  Plasma concentration, ng/mL
Plasma pharmacokinetics of ZE50-0134 with and without rabeprazole (PPI) | Within 60 min prior to dosing with ZE50-0134/placebo to 168 hours post-dose
  To evaluate and compare the PK profile of ZE50-0134 after single dose administration with and without rabeprazole (PPI) pre-dosing in healthy adult volunteers

SECONDARY OUTCOMES:
Safety of ZE50-0134 | From the signing of the consent form until day 8 for all dose levels except level 2 + Itraconazole and until day 11 for dose level 2 + Itraconazole.
  Incidence of AEs/SAEs (serious adverse events)including significant changes from baseline in body weight, vital signs, electrocardiogram parameters and laboratory assessments qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research, Sydney, Randwick NSW, Australia

IPD SHARING:
Plan to Share IPD: No